CLINICAL TRIAL: NCT07225387
Title: Safety and EfficacY of CombinatioN Belimumab and Voclosporin in the TrEatment of PRoliferative Forms of Lupus Glomerulopathy: Synergy Trial
Acronym: SYNERGY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NephroNet, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NephroNet-24-009
Record Dates: First submitted 2025-09-26; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; Voclosporin; Belimumab; MMF; MPA; Prednisone; Proteinura; SYNERGY
MeSH Terms: conditions — Lupus Nephritis | interventions — voclosporin

STUDY DESIGN:
Intervention Model Description: The trial has 2 interventional arms. One treatment regimen is provided to study subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EARLY MMF TERMINATION (90 days) ARM (Active Comparator): EARLY MMF TERMINATION (90 days) ARM in which subjects are randomized 1:1
  Interventions: Drug: Voclosporin
- EXTENDED MMF (360 days) ARM (Active Comparator): EXTENDED MMF TERMINATION (360 days) ARM in which subjects are randomized 1:1
  Interventions: Drug: Voclosporin

INTERVENTIONS:
Drug: Voclosporin — The trial is an open label, parallel, randomized study with patients randomized 1:1 the EARLY MMF TERMINATION (90 days) ARM or the EXTENDED MMF (360 days) ARM looking at the addition of Voclosporin in patients with Lupus Nephritis taking Belimumab, MMF, and Prednisone.

SUMMARY:
This is a Phase IV, open-label, randomized trial to determine whether the combination of Belimumab (BEL) and Voclosporin (VCS), plus background therapy with Mycophenolate Mofetil (MMF), improves the proportion of patients with proliferative lupus nephritis achieving complete renal response (CRR) compared to proportion of patients achieving CRR from recent clinical trials. This protocol will additionally determine whether combination therapy using Belimumab (BEL) and Voclosporin (VCS) facilitates rapid discontinuation of MMF.

DETAILED DESCRIPTION:
Lupus nephritis (LN) is the most serious common manifestation of systemic lupus erythematosus (SLE) and will ultimately affect about half of patients with SLE. LN increases the morbidity and mortality of patients with SLE, especially if Chronic Kidney Disease (CKD) and end-stage kidney disease (ESKD) develop. Morbidity and mortality are significantly mitigated if treatment-induced complete remission (CR) is achieved. While partial remission (PR) is better than no remission, its impact on renal survival is much less than CR. Within the last two years VCS and BEL have been approved for the treatment of LN, bescause each drug was shown to increase the number of patients having CR in well-conducted phase III trials. However, the overall proportion of patients achieving CR was below 50% in each trial, leaving a large unmet need for most patients with LN. Because VCS and BEL target different effector arms of the immune system relevant to kidney injury in LN, and individually have excellent safety profiles, investigators postulated that for the treatment of LN the combination of VCS and BEL with a significant reduction in mycophenolate-based immunosuppression may be complementary and safe, and would ultimately increase the proportion of patients who achieve a CR. In addition, both drugs offer different kidney-protective effects that favor long-term preservation of kidney function. Specifically, VCS protects podocytes and BEL reduces the LN flare rate and through unknown mechanisms, attenuates the decline in GFR seen in LN patients. Investigators further postulate that the combination of these targeted treatments will significantly reduce the need for non-specific immunosuppressives (cytotoxic agents and antimetabolites).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age 18-80 years at time of signing Informed Consent Form
3. Ability to comply with the study protocol, in the investigator's judgment
4. A diagnosis of SLE by any one of the following criteria: European League Against Rheumatism/ American College of Rheumatology/Systemic Lupus International Collaborating Clinics (EULAR/ACR/SLICC)

   • At least one positive ANA defined as a >1:80 titer or a positive anti-ds-DNA within the last 3 years will be accepted.
5. ISN/RPS 2003 Class III, Class IV, Class III/V or Class IV/V Lupus Nephritis diagnosed and meet one of these criteria:

   i) A new diagnosis of LN (kidney biopsy current by SOC), or ii) A previous diagnosis of LN that has been treated, responded, but has flared (If diagnostic biopsy was >24 months before SCREENING, a SOC repeat biopsy will be required for trial entry or by Medical Monitor approval if the last biopsy was less than 36 months prior to screening), or iii) A current diagnosis of LN confirmed by SOC kidney biopsy within the last 24 months prior to screening, or by Medical Monitor approval if the last biopsy - was less than 36 months prior to screening, who has been treated with MMF + glucocorticoids
6. UPCR must be >750 mg/gm from a 24 hour urine collection during screening. If the UPCR does not exceed 750 mg/gm, it may be repeated once during the screening period.
7. Resting systolic blood pressure <150 mm Hg and resting diastolic blood pressure <90 mm Hg.

   Note: If the blood pressure is >150/90 at screening it can be repeated twice in the screening period and if it is <150/90 upon repeat the subject is eligible for study enrollment.
8. Subject must be on maximum tolerated ACEi or ARB therapy as adjudicated by the site PI for ≥4 weeks prior to randomization.

   Note: Patients with confirmed ACEi or ARB intolerance defined as persistent cough, anaphylaxis, or angioedema will be eligible and treatment with another protein-lowering anti-hypertensive encouraged (See #9).
9. Use of other protein-lowering agents, including non-dihydropyridine calcium channel blockers, sodium-glucose transporter 2 (SGLT2) inhibitors, mineralocorticoid receptor antagonists (MRA), will be allowed provided dosing has been stable for ≥4 weeks prior to randomization.

   Note: Titration of the above antihypertensive agents will NOT be allowed following randomization without Sponsor approval. Control for changes in blood pressure will be accomplished using non-protein lowering agents (e.g. Amlodipine, Nifedipine, or Hydralazine).
10. EGFR >30 ml/min/1,73m2 will be required for kidney biopsies obtained >3.0 months from the start of drug administration.

    EGFR> 20 mls/min/1.73 m2 will be allowed for renal biopsies obtained <3.0 months from start of study drug administration provided interstitial fibrosis/tubular atrophy and/or global glomerulosclerosis <65%, and in the judgement of the PI the decrease in eGFR is due to ATN that is reversible.

    Note: All patients will interstitial fibrosis/tubular atrophy and/or global glomerulosclerosis >65% will be excluded from the trial Note: If a patient underwent a renal biopsy within 6 months of randomization and found to have a eGFR between 20-30 ml/min/1,73m2, the site will consult with the study Medical Monitor(s) to determine eligibility.

    Note: The rationale for this is to allow patient to that have low eGFR with intense and active inflammation.
11. Eligible patients will have adequate hematologic parameters defined below as:

    1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
    2. Absolute lymphocyte count (ALC) ≥ 1.0 x 109/L. Note: If count is between .5 x 109/L and 1.0 x 109/L , the site will consult with the study Medical Monitor(s) to determine eligibility.
    3. Platelet count > 75 x 109/L
    4. Hemoglobin > 8.5 g/dL
12. Subjects must be taking Belimumab prior to Consent / Screening or start on Day 0 / Baseline (randomization to short-term MMF or MPA therapy or extended MMF or MPA therapy).

    Note: If Belimumab therapy is expected for less than 12 months in duration post-randomization, please contact Sponsor for approval on a case-by-case basis.
13. Subjects of Child-Bearing Potential must use a highly effective method of contraception consistently and correctly during the study.

Highly effective methods of contraception have a failure rate of <1% per year when used consistently and correctly.

The following methods of contraception are considered highly effective:

* Combined hormonal (estrogen+progestin) contraception (oral, intravaginal, transdermal) associated with inhibition of ovulation.
* Progestogen- or progestin-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation.
* Intrauterine device.
* Intrauterine hormone-releasing system.
* Bilateral tubal ligation/occlusion/division.
* Vasectomized partner (considered a highly effective birth control method provided that partner is the sole sexual partner of the study subject and that the vasectomized partner has received medical assessment of the surgical success).
* Sexual abstinence: defined as refraining from intercourse which may result in pregnancy during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the subject.

Note: Subjects who are on oral contraceptive must also use additional barrier contraceptive methods, consistent with the approved prescribing information for MMF and MPA.

Exclusion Criteria:

1. Currently on renal replacement therapy (dialysis or a kidney transplant), has had dialysis within 3 months of screening or is expected to require renal replacement therapy within 6 months of screening 2. Received cyclophosphamide within 12 weeks of study drug administration 3. Has received treatment with any of the following prior to screening:

a) Rituximab or Obinutuzumab within 24 weeks of screening and there is no measure of circulating C19 B cells. If the measure of circulating C19 B cells is over 10%, the subject will be eligible for study participation.

b) Use of Atacicept, BION-1301, Sibeprenlimab, Povetacicept, or other agents, with the exception of Belimumab, that directly inhibit B call activating factor (BAFF) and/or a proliferation inducing ligand (APRIL) within 12 weeks of study screening.

4. Use of High dose Human Immunoglobulin therapy, abatacept, adalimumab, infliximab, certolizumab, etanercept, golimumab, anakinra, canakinumab, tocilizumab, sarilumab, Satralizumab, Ustekinumab, and Anifrolumab within 12 weeks of study screening.

5. Pure Class V LN on biopsy. 6. In the opinion of the Investigator, subject does not require long-term immunosuppressive treatment (in addition to corticosteroids).

7. Any known hypersensitivity or contraindication to MMF, MPA, Cyclosporine, Tacrolimus, Voclosporin Corticosteroids, Belimumab or any components of these drug products.

8. Current or medical history of:

1. Pancreatitis or gastrointestinal hemorrhage within 6 months prior to screening.
2. Active unhealed peptic ulcer within 3 months prior to screening. If an ulcer has healed and the subject is on adequate therapy, the subject may be randomized. 9. Positive human immunodeficiency virus (HIV) infection. 10. In the opinion of the Investigator, clinically significant drug or alcohol abuse 2 years prior to screening.

   11. Known malignancy within 5 years of screening, with the exception of basal and squamous cell carcinomas of the skin Note: Subjects with cervical dysplasia that is CIN1, but have been treated with conization or LEEP, and have had a normal repeat PAP are allowed.

   12: Lymphoproliferative disease or previous total lymphoid irradiation. 13. Known viral infection (such as HBV and HCV) within 3 months of screening. If HBC and HCV status is unknown, testing should be performed during screening. Subjects with past medical history of HBC or HCV exposure with positive antibodies may be enrolled if a DNA PCR test was negative.

   14. Active tuberculosis (TB), or known history of TB/evidence of old TB if not taking prophylaxis with isoniazid. QuantiFERON gold test must be negative at screening or subject taking isoniazid. Note: If positive at screening the subject can be screen failed, treated, and rescreened in 4 weeks with a confirmed negative chest x-ray.

   15. Patients with known "poor intravenous access" WILL be allowed to participate having placement of a "passport",or port, central IV access or its equivalent for subjects requiring IV infusions of Belimumab upon review and approval by the Medical Monitor 16. Other known clinically significant active medical conditions, such as:

a) Severe cardiovascular disease, including congestive heart failure b) history of cardiac dysrhythmia or congenital long QT syndrome. QTcF (QT interval duration corrected for heart rate using method of Fridericia) exceeding 480 msec in the presence of a normal QRS interval (<110 msec) on historic ECG, if available. An ECG is not is not required for study entry.

17. Liver dysfunction (aspartate aminotransferase, alanine aminotransferase, or bilirubin greater than 2.5 times the upper limit of normal) at screening.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: Day 360 (12 Month) Outcome | 12 months
  Proportion of Patients achieving and maintaining a Complete Clinical Renal Remission (CCRR) at 12 months.
  CCRR is defined as: UPCR≤ 0.5, eGFR≥60 and not >20% below baseline, no rescue meds, sustained on repeat assessment 30 days later.

SECONDARY OUTCOMES:
Secondary Outcome Measure #1: Day 180 (6 Month) Outcome | 6 months
  Proportion of Patients achieving and maintaining a Complete Clinical Renal Remission (CCRR) at 6 months.
  CCRR is defined as: UPCR≤ 0.5, eGFR≥60 and not >20% below baseline, no rescue meds.
Secondary Outcome Measure-#2: | 6 and 12 months
  Proportion of Patients achieving and maintaining a Partial Clinical Renal Remission (PCRR) at 6 and 12 months.
  PCRR is defined as: A UPCR from a SPOT or 24-hour urine collection ≤50% of UPCR at baseline and eGFR not >20% below baseline eGFR sustained on repeat measurement at Day 180 (6 months) and Day 360 (12 months).
Secondary Outcome Measure-#3: | 12 months
  Effectiveness of combination therapy on successful discontinuance of MMF. Examine the proportion of patients achieving CCRR who discontinued MMF after 90 days and compare to the proportion of patients achieving CCRR who continued MMF for the 360 Day (12 month) duration of the trial. Expectation is no difference in efficacy.
Secondary Outcome Measure-#4: | 12 months
  The proportion of patients requiring rescue therapy. Rescue therapy defined as: A patient requiring an increase in glucocorticoid (prednisone) to 1 mg/kg/d or intravenous solumedrol >80 mg for over a week, or the addition of, or change to cyclophosphamide, eculizumab, rituximab, therapeutic plasmapheresis, or an experimental therapeutic.

CONTACTS AND LOCATIONS:
Overall Officials: James Tumlin, MD, Principal Investigator — NephroNet, Inc.
Locations (7):
- United States (7):
  - AARA Clinical Research, Glendale, Arizona
  - Piedmont Physicians Rheumatology, Atlanta, Georgia
  - Georgia Nephrology Research Institute, Lawrenceville, Georgia
  - Parris & Associates, Lawrenceville, Georgia
  - Nephrology Clinical Trials Unit The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - AARA Clinical Research, Fort Worth, Texas